CLINICAL TRIAL: NCT03452826
Title: Combined Use of a Respiratory Broad Panel MULTIplex PCR and Procalcitonin to Reduce Antibiotics Exposure in Patients With Severe Community-Acquired Pneumonia: a Multicentre, Parallel-group, Open-label, Randomized Controlled Trial.
Brief Title: Combined Use of a Respiratory Broad Panel mPCR and Procalcitonin to Reduce Duration of Antibiotics Exposure in Patients With Severe Community-Acquired Pneumonia
Acronym: MULTI-CAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P160928J; AO 1615-48 (Other Grant/Funding Number: PHRC)
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Community-acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antibiotic therapy according to the result of mPCR (Experimental): Combined use of a respiratory broad panel Multiplex polymerase chain reaction (mPCR) (performed on a lower respiratory tract sample : bronchoalveolar lavage fluid or tracheal aspirate, otherwise sputum) and procalcitonin.
  Interventions: Device: Antibiotic therapy according to the result of mPCR (device)
- Antibiotic therapy at discretion of ICU physicians (No Intervention): Antibiotic therapy at discretion of ICU physicians

INTERVENTIONS:
Device: Antibiotic therapy according to the result of mPCR (device) — * Phone call at D28 and D90, unless the patient is still hospitalized;
  * Collection of a respiratory tract sample (either distal, i.e. tracheal aspirate or bronchoalveolar lavage, or proximal, i.e. sputum) for broad panel respiratory mPCR in the intervention arm.
  * Collection of an additional respiratory tract sample for biological banking in both arms.
  Other Names: Antibiotic therapy to be adapted according to the result of mPCR (device)
  Arms: Antibiotic therapy according to the result of mPCR

SUMMARY:
To assess the effectiveness of a management strategy combining a broad panel respiratory mPCR and an algorithm of early antibiotic de-escalation and discontinuation based on both the mPCR results and the procalcitonin (intervention) in severe CAP, as compared to a conventional strategy (control).

A multicentre, parallel-group, open-label, randomized controlled trial. The primary assessment criterion est the number of antibiotic-free days at 28 days

DETAILED DESCRIPTION:
Randomization is performed immediately after the inclusion.

* In the intervention arm, a broad panel respiratory mPCR is performed on a lower respiratory tract sample (bronchoalveolar lavage fluid or tracheal aspirate, otherwise sputum), collected before the 12th hour following inclusion.
* In both arms, an additional lower respiratory tract sample (bronchoalveolar lavage fluid or tracheal aspirate, otherwise sputum) is collected for biological studies and banking.
* In the intervention arm, an algorithm of early antibiotic de-escalation and discontinuation is based on the early microbiological results, including the mPCR results, and the procalcitonin value. This algorithm is applied as soon as possible (before the 24th hour following inclusion if possible).
* In the control arm, initial antibiotic therapy is maintained, according to guidelines.
* In both arms, after 72 hours of antibiotic therapy, ICU physicians are advised to use procalcitonin (values and kinetics) to guide antibiotic therapy discontinuation, with a recommended total duration of 7 days, unless otherwise indicated.
* In both arms, a switch to oral therapy is encouraged

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) with CAP admitted to the ICU since 18 hours or less; the diagnosis of pneumonia includes two clinical criteria among a temperature > 37.8°C, tachypnea (respiratory rate > 25/min), chest pain, cough, expectoration, localized crackles, with or without signs of pleural effusion, pulse oximetry less than 92% while breathing room air, and a newly-appeared parenchymal infiltrate; the pneumonia is community-acquired if the time between hospital admission and ICU referral is below or equal to 48 hours.
* Informed consent or emergency procedure.

Exclusion Criteria:

* Pregnancy;
* Congenital immunodeficiency;
* HIV infection with the lymphocyte CD4 count below 200/mm3 or unknown in the last year;
* Acute hematologic malignancy;
* Neutropenia (<1 leucocyte/mL or < 0.5 neutrophil/mL);
* Immunosuppressive drugs within the previous 30 days, including anti-cancer chemotherapy and anti-rejection drugs for organ/bone marrow transplant
* Corticosteroids ≥ 20 mg/d of prednisone equivalent for more than 14 days;
* chronic obstructive pulmonary disease (COPD) with previous history of colonization/infection with Pseudomonas aeruginosa;
* Tracheostomy;
* Diffuse bronchiectasis, cystic fibrosis;
* Aspiration pneumonia;
* Moribund patient or death expected from underlying disease during the current admission;
* Patient deprived of liberty or under legal protection measure;
* Participation in another interventional trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 411 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
The effectiveness of a management combining a broad panel respiratory mPCR and an algorithm of early antibiotic de-escalation and discontinuation based on both the mPCR results and the procalcitonin in severe CAP, as compared to a conventional strategy | Day 28
  the number of antibiotic free days at D28, which corresponds to the number of days alive without any at Day 28.

SECONDARY OUTCOMES:
Mortality at 28 (D28) and 90 days (D90); | Day 28 and day 90
  Mortality rate at D28 and D90
Number of defined daily dose (DDD) per 100 patient days of broad- and narrow-spectrum antibiotics | Day 28
  Number of defined daily dose (DDD) per 100 patient days of broad- and narrow-spectrum antibiotics
Antibiotics duration at D28 | Day 28
  Antibiotics duration at D28
Number of organ-failure free days (based on SOFA) at D28 | Day 28
  Number of organ-failure free days (based on SOFA) at D28
Incidence rates of bacterial superinfections at D28 | Day 28
  Incidence rates of bacterial superinfections at D28
Incidence rates of colonization/infection with multidrug resistant bacteria and Clostridium difficile infections at D28 | Day 28
  Incidence rates of colonization/infection with multidrug resistant bacteria and Clostridium difficile infections at D28
Incidence rates of relapse (same pathogen) or reinfection (another pathogen) at D28 | Day 28
  Incidence rates of relapse (same pathogen) or reinfection (another pathogen) at D28
Duration of ICU and hospital stay | Day 90
  Duration of ICU and hospital stay
Cost of the total hospital admissions (including 90-day repeated admissions), ICU costs, cost of the microbiological diagnostic workup; | Day 90
  Cost of the total hospital admissions (including 90-day repeated admissions), ICU costs, cost of the microbiological diagnostic workup;
Incremental / decremental cost effectiveness ratio in cost per treatment success (90-day composite of all-cause death and infection recurrence). | Day 90
  Incremental / decremental cost effectiveness ratio in cost per treatment success (90-day composite of all-cause death and infection recurrence).
Sensitivity, specificity, and likelihood ratios of the broad panel mPCR Film Array for the diagnosis of pneumonia, taking the conventional microbiological tests as reference | Day 28
  Sensitivity, specificity, and likelihood ratios of the broad panel mPCR Film Array for the diagnosis of pneumonia, taking the conventional microbiological tests as reference
Euroquol questionary (EQ-5D-3L) | Day 90
  Euroquol questionary (EQ-5D-3L)
To assess the operational values of the broad panel mPCR Film Array for the diagnosis of ventilator associated pneumonia (in the intervention group only). | Day 28
  Sensitivity, specificity, and likelihood ratios of the broad panel mPCR Film Array for the diagnosis of ventilator associated pneumonia (in the intervention group only), taking the conventional microbiological tests as reference.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François TIMSIT, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital BICHAT, Paris, France

REFERENCES:
- [Derived] Voiriot G, Argaud L, Cohen Y, Tuffet S, Chauvelot L, Souweine B, Klouche K, Reignier J, Schwebel C, Rouze A, Mekontso Dessap A, Bohe J, Megarbane B, Carvelli J, Navellou JC, Gibot S, Maury E, Dellamonica J, Dequin PF, Dessajan J, Armand-Lefevre L, Vandenesch F, Verdet C, Durand Zaleski I, Berard L, Rousseau A, Tabassome S, Fartoukh M, Timsit JF; MULTI-CAP collaborative trial group. Combined use of a multiplex PCR and serum procalcitonin to reduce antibiotic exposure in critically ill patients with community-acquired pneumonia: the MULTI-CAP randomized controlled trial. Intensive Care Med. 2025 Aug;51(8):1417-1430. doi: 10.1007/s00134-025-08014-9. Epub 2025 Jul 15. PMID 40663137
- [Derived] Voiriot G, Fartoukh M, Durand-Zaleski I, Berard L, Rousseau A, Armand-Lefevre L, Verdet C, Argaud L, Klouche K, Megarbane B, Patrier J, Richard JC, Reignier J, Schwebel C, Souweine B, Tandjaoui-Lambiotte Y, Simon T, Timsit JF; MULTI-CAP study group. Combined use of a broad-panel respiratory multiplex PCR and procalcitonin to reduce duration of antibiotics exposure in patients with severe community-acquired pneumonia (MULTI-CAP): a multicentre, parallel-group, open-label, individual randomised trial conducted in French intensive care units. BMJ Open. 2021 Aug 18;11(8):e048187. doi: 10.1136/bmjopen-2020-048187. PMID 34408046
- [Derived] Kerneis S, Visseaux B, Armand-Lefevre L, Timsit JF. Molecular diagnostic methods for pneumonia: how can they be applied in practice? Curr Opin Infect Dis. 2021 Apr 1;34(2):118-125. doi: 10.1097/QCO.0000000000000713. PMID 33395094